CLINICAL TRIAL: NCT03043976
Title: Using Step Count to Enhance Daily Physical Activity in Pulmonary Hypertension
Acronym: STEPinPH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated early due to ligistic reasons with study staff
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15/LO/1185
Record Dates: First submitted 2016-09-09; First posted 2017-02-06 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Hypertension, Pulmonary
Keywords: Physical activity; Steps count
MeSH Terms: conditions — Hypertension, Pulmonary; Motor Activity

STUDY DESIGN:
Intervention Model Description: Partial crossover. A group of 10 underwent the intervention, a group of 10 was observed for 8 weeks without receiveng any feedback, then underwent the intervention. The main outcome was evaluated as the difference between the end of intervention and baseline (paired data). We did not recuit any patient in arm 3.
Oversight: Data Monitoring Committee: No

ARMS (3):
- feedback and goal-setting group (Active Comparator): At the baseline, patients will fill a questionnaire about their quality of life (SF36), will perform a 6'walk test (6MWT), will undertake a blood sample (BNP). In the run-in period (1 week) patients will wear an Actigraph GT9X Link device which only displays the time and the battery level; all activity data will be recorded. Then participants will wear an Actigraph GT9X Link device which shows real time data about the number of steps and will upload their data via the Study Admin Mobile application for smartphones/tablets. Patients will be asked to aim for an average specified number of steps/day week by week and will receive a weekly report with results from the previous week and targets to achieve. After 8 weeks, patients will attend visit 2 (6MWT, SF36 and BNP assessment) and will carry on wearing the activated device for 8 weeks receiving weekly feedbacks and targets. After 8 weeks patients will attend visit 3 (6MWD, SF36 and BNP will be assessed) which is the end of the study.
  Interventions: Device: Actigraph GT9X Link device
- Control group (Active Comparator): At the baseline, patients will fill a questionnaire about their quality of life (SF36), will perform a 6'WT and will undertake a blood sample (BNP). After a run-in period (1 week) with an Actigraph GT9X Link device disabled from showing the number of steps, patients will wear an Actigraph GT9X Link device which still only displays time and battery level and will upload data via the Study Admin Mobile application for smartphones/tablets without receiving any feedback. After 8 weeks, patients will be assessed (SF36, 6'WT, BNP) and will start to wear a new device enabled to display the daily step count. Patients will be asked to aim for an average specified number of steps/day, receiving a weekly summary of the previous week with targets to achieve week by week. After 8 weeks, patients will be assessed (6'WT, SF36, BNP) and will carry on wearing the device and receiving feedbacks and targets for a further 8 week period, after that patients will be finally assessed (SF36, 6'WT, BNP)
  Interventions: Device: Actigraph GT9X Link device
- newly diagnosed patients (Placebo Comparator): In the week leading up to their inpatient admission for diagnostic investigations, patients who are treatment-naïve will be given the Actigraph GT9X Link device which will only display the time and the charge level of the battery. Patients will be asked, as well, to fill a questionnaire about their quality of life, to perform a 6MWT and a blood sample (BNP). As soon as patients start the drug therapy, patients will wear a second Actigraph GT9X Link device still disabled from showing real time data about the number of daily steps. Participants will not receive any feedback during the whole period and will be asked, as well, to upload the data collected through the remote mobile system. At their first clinical assessment (after about 4 or 5 weeks), 6'WT, BNP and questionnaire about quality of life will be reassessed.
  If patients are not being started on drug therapy then they will be withdrawn from the study
  Interventions: Device: Actigraph GT9X Link device

INTERVENTIONS:
Device: Actigraph GT9X Link device — Assessment of the level of physical activity of PH patients using the Actigraph GT9X Link device that includes a triaxial accelerometer and can be enabled to show on its display the number of steps taken for the day, so that it can also be used by the patients as a common pedometer.
  Evaluation of the effects of an 8 week step count-based light touch training programme to see if activity can be increased

SUMMARY:
This study will collect information about physical activity in patients affected by pulmonary hypertension, through a specific device that can be worn on the wrist, and which measures daily step count. The purpose of the study is to demonstrate whether providing patients with their daily step count can increase their levels of daily activity if they have some basic targets to achieve. Investigators also wish to compare the effects of this approach in increasing daily physical activity, with the benefit gained when a drug therapy for pulmonary hypertension is initiated, in patients that have just been diagnosed.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a rare and progressive disorder and shortness of breath and fatigue, especially during exercise, are very common symptoms, resulting in a reduced capacity to perform daily activities and in an impaired quality of life. Furthermore, reduced exercise capacity in PH is associated with depression and anxiety disorders. Recent literature reveals a strong association of sedentary time with adverse cardiovascular outcomes, so that the development of therapeutic strategies to avoid this event is pivotal in the management of PH, in addition to the beneficial results of modern medical treatment. Recently the role of exercise and rehabilitation in different respiratory and cardiac conditions has been evaluated in the literature, overtaking the concerns raised in the past that exercise could worsen the condition and thus the progression of these kind of diseases, but just a few studies have been done in patients affected by PH.

International guidelines on pulmonary hypertension recommend avoiding strenuous exercise that leads to distressing symptoms, while encourage low level graded aerobic exercise, such as walking, as tolerated. Nonetheless, little is still known about the effects of lifestyle changes, such as the amount of physical activity that patients can or should practice. Pedometers have been used to enhance the daily physical activity and to improve, when assessed, some prognosis related outcomes, both in healthy subjects and those affected by different pathological conditions, in particular cardiac and respiratory diseases. However, a training model based on step count targets has never been evaluated in PH, to our knowledge. Step counting devices have recently experienced a surge in popularity as a tool for motivating and monitoring physical activity in the general population, especially combined with applications for smartphones, that provide feedback, such as an overview of the data recorded. Thus, it seems reasonable to explore the opportunity to develop a step count based training model to enhance daily exercise in PH patients, through these non-invasive, patient friendly and relatively inexpensive devices.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Nice Classification Groups 1 and 4 Pulmonary Hypertension (pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension)
* WHO functional class I-IV
* Stable on current medication for 8/52 for group 1 (feedback and goal-setting group) and group 2 (control group)
* For group 3 (newly diagnosed patients), treatment-naïve patients undergoing investigation who are likely to start therapy (based on clinical judgment of the clinician)
* Patients with handheld devices (such as smartphones or tablets) which can run the Study Admin Mobile application.

Exclusion Criteria:

* Pregnancy: we will screen for this on the basis of the history from the patient, and if she is not sure if she might be pregnant, a pregnancy test will be offered
* Malignant arrhythmias
* Syncope within the last 6 months
* Skeletal or muscle abnormalities prohibiting walking

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in daily physical activity | From baseline to 16 - 25 weeks
  The principal objective is to demonstrate a difference in the intensity of daily physical activity, measured in activity counts per minute, from the basal period to the last week of the 8-week training programme compared with control

SECONDARY OUTCOMES:
Change in 6MWT | From baseline to 16 - 25 weeks
  Evaluation of the difference in the 6MWT from the basal period to the end of the 8-week training programme compared with control
Change in BNP | From baseline to 16 - 25 weeks
  Evaluation of the difference in BNP values from the basal period to the end of the 8-week training programme compared with control
Change in Quality of life | From baseline to 16 - 25 weeks
  Evaluation of the difference in quality of life (assessed by SF36 questionnaire) from the basal period to the end of the 8-week training programme compared with control
Long-term effects of training protocol | End of the 8 week period
  Evaluate if the eventual benefit gained after the 8 week training period (measured in activity counts per minute) is maintained, reduced or increased for a further 8 week period (group1+ group 2).
Comparison between training protocol and initiation of PH treatment in terms of increased physical activity | 5-6 weeks
  Comparing the efficacy of our training protocol to the effects of the initiation of the PH drug treatment in newly diagnosed patients, in terms of increased physical activity assessed in terms of activity counts.

CONTACTS AND LOCATIONS:
Overall Officials: Luke SGE Howard, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Background] Grunig E, Lichtblau M, Ehlken N, Ghofrani HA, Reichenberger F, Staehler G, Halank M, Fischer C, Seyfarth HJ, Klose H, Meyer A, Sorichter S, Wilkens H, Rosenkranz S, Opitz C, Leuchte H, Karger G, Speich R, Nagel C. Safety and efficacy of exercise training in various forms of pulmonary hypertension. Eur Respir J. 2012 Jul;40(1):84-92. doi: 10.1183/09031936.00123711. Epub 2012 Feb 9. PMID 22323570
- [Background] Mainguy V, Provencher S, Maltais F, Malenfant S, Saey D. Assessment of daily life physical activities in pulmonary arterial hypertension. PLoS One. 2011;6(11):e27993. doi: 10.1371/journal.pone.0027993. Epub 2011 Nov 16. PMID 22110770
- [Background] de Man FS, Handoko ML, Groepenhoff H, van 't Hul AJ, Abbink J, Koppers RJ, Grotjohan HP, Twisk JW, Bogaard HJ, Boonstra A, Postmus PE, Westerhof N, van der Laarse WJ, Vonk-Noordegraaf A. Effects of exercise training in patients with idiopathic pulmonary arterial hypertension. Eur Respir J. 2009 Sep;34(3):669-75. doi: 10.1183/09031936.00027909. PMID 19720810
- [Background] Mendoza L, Horta P, Espinoza J, Aguilera M, Balmaceda N, Castro A, Ruiz M, Diaz O, Hopkinson NS. Pedometers to enhance physical activity in COPD: a randomised controlled trial. Eur Respir J. 2015 Feb;45(2):347-54. doi: 10.1183/09031936.00084514. Epub 2014 Sep 26. PMID 25261324
- [Background] McLaughlin VV, Archer SL, Badesch DB, Barst RJ, Farber HW, Lindner JR, Mathier MA, McGoon MD, Park MH, Rosenson RS, Rubin LJ, Tapson VF, Varga J, Harrington RA, Anderson JL, Bates ER, Bridges CR, Eisenberg MJ, Ferrari VA, Grines CL, Hlatky MA, Jacobs AK, Kaul S, Lichtenberg RC, Lindner JR, Moliterno DJ, Mukherjee D, Pohost GM, Rosenson RS, Schofield RS, Shubrooks SJ, Stein JH, Tracy CM, Weitz HH, Wesley DJ; ACCF/AHA. ACCF/AHA 2009 expert consensus document on pulmonary hypertension: a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents and the American Heart Association: developed in collaboration with the American College of Chest Physicians, American Thoracic Society, Inc., and the Pulmonary Hypertension Association. Circulation. 2009 Apr 28;119(16):2250-94. doi: 10.1161/CIRCULATIONAHA.109.192230. Epub 2009 Mar 30. No abstract available. PMID 19332472
- [Background] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Background] Pugh ME, Buchowski MS, Robbins IM, Newman JH, Hemnes AR. Physical activity limitation as measured by accelerometry in pulmonary arterial hypertension. Chest. 2012 Dec;142(6):1391-1398. doi: 10.1378/chest.12-0150. PMID 22576635
- [Background] Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G; ESC Committee for Practice Guidelines (CPG). Guidelines for the diagnosis and treatment of pulmonary hypertension: the Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS), endorsed by the International Society of Heart and Lung Transplantation (ISHLT). Eur Heart J. 2009 Oct;30(20):2493-537. doi: 10.1093/eurheartj/ehp297. Epub 2009 Aug 27. No abstract available. PMID 19713419
- [Background] Ulrich S, Fischler M, Speich R, Bloch KE. Wrist actigraphy predicts outcome in patients with pulmonary hypertension. Respiration. 2013;86(1):45-51. doi: 10.1159/000342351. Epub 2012 Dec 11. PMID 23234873